CLINICAL TRIAL: NCT03549221
Title: Efficacy of Adrenaline in Periarticular Analgesic Injection on Postoperative Pain Control After Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Efficacy of Adrenaline in Periarticular Analgesic Injection on Postoperative Pain Control After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaturong Pornrattanamaneewong, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 696/2560
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
Keywords: total knee arthroplasty; multimodal anesthetic cocktail; adrenaline; morphine consumption; blood loss; Levobupivacaine
MeSH Terms: conditions — Pain, Postoperative; Hemorrhage | interventions — Epinephrine; Levobupivacaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAC with adrenaline (Experimental): the multimodal anesthetic cocktail (MAC) consisted of 100 mg Levobupivacaine (0.5%, 20 mL) 30 mg ketorolac (1 ml) and 0.6 mg 1:1000 epinephrine (0.6 ml). They were mixed with a 0.9% normal saline solution to a total volume of 100 ml.
  Interventions: Drug: 0.6 mg 1:1000 epinephrine (0.6 ml)
- MAC without adrenaline (No Intervention): the multimodal anesthetic cocktail (MAC) consisted of 100 mg Levobupivacaine (0.5%, 20 mL) and 30 mg ketorolac (1 ml). They were mixed with a 0.9% normal saline solution to a total volume of 100 ml.

INTERVENTIONS:
Drug: 0.6 mg 1:1000 epinephrine (0.6 ml) — In group 1, the multimodal anesthetic cocktail consisted of 100 mg Levobupivacaine (0.5%, 20 mL) 30 mg ketorolac (1 ml) and 0.6 mg 1:1000 epinephrine (0.6 ml). In group 2, the multimodal anesthetic cocktail consisted of 100 mg Levobupivacaine (0.5%, 20 mL) and 30 mg ketorolac (1 ml). Both groups were mixed with a 0.9% normal saline solution to a total volume of 100 ml.
  Other Names: 100 mg Levobupivacaine (0.5%, 20 mL); 30 mg ketorolac (1 ml)
  Arms: MAC with adrenaline

SUMMARY:
Multimodal anesthetic drug injection has been used extensively and the results of many studies suggest that postoperative pain can relief and improve the postoperative satisfaction of patients. Adrenaline is a combination of multimodal anesthetic cocktail to relieve pain. It is believed that Adrenaline causes vasoconstriction, reduces absorption of anesthetic drug into the system circulation. Currently, a comparative study on the effect of pain reduction of Adrenaline injection in the anesthetic cocktail is relatively low. There are different doses in each institution. In addition, the use of new anesthetic is Levobupivacaine that has more vasoconstrictive effect compare with traditional Bupivacaine. It also reduces the side effects of systemic and cardiotoxic effect. Therefore, the investigators think that It may not be necessary to mix Adrenaline in the multimodal anesthetic drug. Levobupivacaine already to avoid the potential side effects of Adrenaline.

DETAILED DESCRIPTION:
The patients will be divided into two groups. In group 1, the multimodal anesthetic cocktail consisted of 100 mg Levobupivacaine (0.5%, 20 mL) and 30 mg ketorolac (1 ml). In group 2, the multimodal anesthetic cocktail consisted of 100 mg Levobupivacaine (0.5%, 20 mL), 30 mg ketorolac (1 ml) and 0.6 mg 1:1000 epinephrine (0.6 ml). Both groups were mixed with a 0.9% normal saline solution to a total volume of 100 ml. The outcome research assistant who collects data was blinded to the treatment groups. Patients will be treated with the routine standard regimen for total knee arthroplasty. Surgeons will use same surgical techniques through a standard medial parapatellar approach. In addition, standardized posterior-stabilized TKA (Zimmer Nexgen LPS flex) was used in all patients. After bone cutting before inserting the actual implant, the assistant scrub nurse in the operating room will open the envelope that the patient was classified in group 1 or group 2 and perform mixing according to the prescribed medication. The doctor who undergoes surgery was blinded. The anesthetic cocktail was divided into 4 parts 25 ml each and it was injected into 4 areas. First 25 ml cocktail was injected into the posterior capsule (P), posteromedial (PM) and posterolateral capsule (PL). The second part was injected into the medial gutter (M). The third part was injected into the lateral gutter and the forth part was injected into quadriceps muscle, retinacula tissues, pes anserinus, suprapatellar and infrapatellar fat pads (A). During the first 48 hours, all patients received intravenous morphine prn for pain, as well as dynastat, Tylenol with codeine, as required, for control of pain. After 48 hours, the pain was controlled by oral intravenous morphine and medication as requires until the patient was discharged from the hospital.

The primary outcome measure was the severity of postoperative pain during the first 48 hours after surgery. The pain was assessed by a Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (extreme pain) every 6 hours postoperatively. Secondary outcome measures compared the consumption of intravenous morphine, which was measured every six hours in 48 hours after surgery. Additionally, blood loss in the drain at 24, 48 hours was recorded. Any complications following surgery were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee osteoarthritis
* Aged between 40 and 80 years
* Must be able to understand and willing to follow instructions

Exclusion Criteria:

* Patients unable to undergo anesthesia during surgery by spinal block or adductor block
* Patients with the history of levobupivacaine, etoricoxib drug allergy
* Patients with the history of allergic or nausea vomiting severely when receiving morphine
* Patients with kidney disease who have a creatinine clearance of less than 50 ml/min, cirrhosis, cardiovascular disease, stroke, poorly controlled hypertension
* Patients with the history of venous thrombosis
* Patients with complications during surgery such as torn ligaments
* Patients who refuse to participate in the research.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
the severity of postoperative pain | The first 48 hours after surgery
  The pain was assessed by a Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (extreme pain) every 6 hours postoperatively.

SECONDARY OUTCOMES:
the consumption of intravenous morphine | The first 48 hours after surgery
  the consumption of intravenous morphine, which was measured every six hours
blood loss in the drain | at 24, 48 hours after surgery
  blood loss in the radivac drain

CONTACTS AND LOCATIONS:
Overall Officials: Keerati Chareancholvanich, MD, Study Chair — Mahidol University
Locations (1):
- Chaturong Pornrattanamaneewong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No